CLINICAL TRIAL: NCT06914960
Title: Ultrasound-Guided Genicular Nerve Radiofrequency Ablation Therapy: Effectiveness of 5 Nerve Protocols Versus 3 Nerve and 2 Nerve Protocols - A Prospective Randomized Controlled Study
Brief Title: Efficacy of Ultrasound-Guided Genicular Nerve Radiofrequency Ablation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bengu Turemenogullari (Other Government)
Responsible Party: Sponsor-Investigator, Bengu Turemenogullari, Principal Investigator, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Genicular nerve RF
Record Dates: First submitted 2025-01-12; First posted 2025-04-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Gonarthrosis
Keywords: gonarthrosis; genicular nerve; radiofrequency; ablation; proprioception; balance; risk of falling; chronic pain
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients and care provider, the physician performing the assessment and the physiotherapist treating the patient will be blind to what procedure is being performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Radiofrequency Ablation Targeting Two Genicular Nerves (Active Comparator): 2 nerve radiofrequency ablation: Superior Medial (SM) and Inferior Medial (IM) branches.
  A group of patients will receive a single treatment session using the Radiofrequency Ablation method for 2 nerves, Superior Medial (SM) and Inferior Medial (IM).
  Interventions: Procedure: 2-point Radiofrequency Ablation
- Radiofrequency Ablation Targeting Three Genicular Nerves (Active Comparator): 3 nerve radiofrequency ablation: Superior Medial (SM), Superıor Lateral (SL) and Inferior Medial (IM) branches.
  A group of patients will receive a single treatment session using the Radiofrequency Ablation method for 3 nerves, Superior Medial (SM), Superior Lateral (SL) and Inferior Medial (IM).
  Interventions: Procedure: 3-point Radiofrequency Ablation
- Radiofrequency Ablation Targeting Five Genicular Nerves (Active Comparator): 5 nerve radiofrequency ablation: Superior Medial (SM), Superıor Lateral (SL), Inferior Medial(IM), Rekurren Fibular Nerve (RFN) and İnfrapatellar Branch of Saphenous Nerve (IPBSN).
  Another group of patients will receive a single treatment session with Radiofrequency Ablation for 5 nerves: Superior Medial (SM), Superior Lateral (SL), Inferior Medial (IM), Recurrent Fibular Nerve (RFN) and Infrapatellar Branch of Saphenous Nerve (IPBSN).
  Interventions: Procedure: 5-point Radiofrequency Ablation

INTERVENTIONS:
Procedure: 2-point Radiofrequency Ablation — For the radiofrequency ablation (RFA) procedure, a 10 cm long, 22 gauge RF cannula with a 10 mm active tip (Model SC-K, Top Neuropole, MPS Medical Product Service GmbH, Germany) will be used.
  In order to increase the accuracy of the location determined by ultrasound, sensory stimulation will be applied at a frequency of 50 Hz and with a threshold value lower than 0.6 volts. In order to prevent the motor nerves from being affected, the absence of lower extremity muscle fasciculations in the relevant area will be confirmed with 2 volt stimulation at 2 Hz frequency. Patients in 2 nerve groups (SM and IM) will undergo 2-point RFA at 42°C using a 120-second pulse RFA generator (TOP Lesion Generator TLG-20, MPS Medical Product Service GmbH, Germany).
  To address any discomfort that may occur after the procedure, a total of 2 cc of betamethasone (5 mg+2 mg/1 cc) and %2 lidocaine (1 cc) will be injected into the points where RFA is applied, after aspiration.
  Arms: Radiofrequency Ablation Targeting Two Genicular Nerves
Procedure: 3-point Radiofrequency Ablation — Description: For the radiofrequency ablation (RFA) procedure, a 10 cm long, 22 gauge RF cannula with a 10 mm active tip (Model SC-K, Top Neuropole, MPS Medical Product Service GmbH, Germany) will be used. In order to increase the accuracy of the location determined by ultrasound, sensory stimulation will be applied at a frequency of 50 Hz and with a threshold value lower than 0.6 volts. In order to prevent the motor nerves from being affected, the absence of lower extremity muscle fasciculations in the relevant area will be confirmed with 2 volt stimulation at 2 Hz frequency. 3-point RFA will be applied to patients in 3 nerve groups (SM, SL and IM) using a generator (TOP Lesion Generator TLG-20, MPS Medical Product Service GmbH, Germany) in the form of 120-second pulse RFA at 42°C. To address any discomfort that may occur after the procedure, a total of 2 cc of betamethasone (5 mg+2 mg/1 cc) and %2 lidocaine (1cc) will be injected into the points where RFA is applied, after aspiration.
  Arms: Radiofrequency Ablation Targeting Three Genicular Nerves
Procedure: 5-point Radiofrequency Ablation — Description: For the radiofrequency ablation (RFA) procedure, a 10 cm long, 22 gauge RF cannula with a 10 mm active tip (Model SC-K, Top Neuropole, MPS Medical Product Service GmbH, Germany) will be used. In order to increase the accuracy of the location determined by ultrasound, sensory stimulation will be applied at a frequency of 50 Hz and with a threshold value lower than 0.6 volts. In order to prevent the motor nerves from being affected, the absence of lower extremity muscle fasciculations in the relevant area will be confirmed with 2 volt stimulation at 2 Hz frequency. 5-point RFA will be applied to patients in 5 nerve groups (SM, SL and IM, recurrent fibular nerve-RFN, infrapatellar branch of saphenous nerve-IPBSN) via same generator in the form of 120-second pulse RFA at 42°C. To address any discomfort that may occur after the procedure, a total of 2cc of betamethasone (5mg+2mg/1cc) and %2 lidocaine (1cc) will be injected into the points where RFA is applied, after aspiration.
  Arms: Radiofrequency Ablation Targeting Five Genicular Nerves

SUMMARY:
The main symptom of knee osteoarthritis, which occurs after damage to the joint cartilage with age, is pain, but this symptom often becomes chronic. Current conservative treatments have moderate effects on chronic knee pain and their use is limited due to the risk of side effects. In addition to pain, patients also experience other symptoms.

As a result of the osteoarthritis process, prorioception in the knee is impaired with a decrease in mechanoreceptors, resulting in loss of balance and an increase in the risk of falling.

DETAILED DESCRIPTION:
Our aim in this study is; to investigate the superiority and long-term effectiveness of radiofrequency ablation therapy applied with 5 nerves, 3 nerves and 2 nerves on fall risk, balance, proprioception, chronic pain and symptoms in knee osteoarthritis.

Radiofrequency ablation therapy; it is effective in chronic pain by causing nerve damage. Application of radiofrequency ablation therapy on chronic knee pain with different protocols has been reported in the literature with different results.

In the literature, it has been shown that the 5-nerve protocol versus the 3-nerve protocol with the radiofrequency ablation method reduces pain and provides functional improvement in patients with chronic knee osteoarthritis. In another study in the literature, functional and physical performance was examined with a 3-nerve protocol in the same patient group without a control group and was found effective.

To our knowledge, there is no study in the literature evaluating the effectiveness of radiofrequency ablation therapy on fall risk, balance and proprioception after applying different protocols in knee osteoarthritis.

There are few studies in the literature regarding radiofrequency ablation treatment procedures for knee osteoarthritis. In line with this information, it is obvious that more studies are needed on the radiofrequency ablation method. Although this method has been shown to be effective and popular in recent years, since it is an invasive procedure, another aim of ours is to reveal what is the least intervention that will give the most effective results for patients.

Diagnostic genicular nerve block: It will be performed by injecting lidocaine (%2, 2 cc) into the superıor lateral (SL), superıor medial (SM) and inferior medial (IM) branches of the genicular nerve passing through the periosteal areas connecting the femoral shaft to the bilateral epicondyles and the tibia shaft to the medial epicondyle.

All patients who meet the study eligibility criteria will undergo a diagnostic genicular nerve block before the procedure, and patients with a decrease in VAS (visual analog scale) of more than 50 percent for more than 24 hours will be considered for the RFA procedure. Injection will be performed under ultrasound guidance using a 12 Mhz linear array transducer probe (GE Logiq P9, GE Healthcare, Boston, MA).

The patients are randomly divided into 3 groups with the help of a computer-based randomization program. One group will be treated with the RFA method for 2 nerves (SM, IM), the other group will be treated with 3 nerves (SM, SL, IM), and the other group will be treated with a single treatment session for 5 nerves (SM, SL, IM, Rekurrent fibular nerve-RFN, Infrapatellar branch of saphenous nerve-IPBSN).

Before the RFA procedure, all participants will be anesthetized with 1 cc %1 lidocaine under sterile conditions, in a supine position, with a pillow placed under the popliteal fossa, and the skin and subcutaneous tissues on the surface of the targeted nerves.

RFA application sites will be determined by finding the arteries between the shaft and epicondyles of the femur and tibia with the help of Color Doppler Ultrasound. The infrapatellar branch of the saphenous nerve (IPBSN) will be confirmed by Doppler Ultrasound of the artery of the nerve 4 cm medial to the apex of the patella and tibial tubercle. Recurrent fibular nerve (RFN) will be confirmed by Doppler Ultrasound of the nerve artery along the caudate line of Gerdy's tubercle, 1 cm below the tuberosity tibia. For the RFA procedure, a 10 cm long, 22 gauge RF cannula with a 10 mm active tip (Model SC-K, Top Neuropole, MPS Medical Product Service GmbH, Germany) will be used.

In order to increase the accuracy of the location determined by ultrasound, sensory stimulation will be applied at a frequency of 50 Hz and with a threshold value lower than 0.6 volts. In order to prevent the motor nerves from being affected, the absence of lower extremity muscle fasciculations in the relevant area will be confirmed with 2 volt stimulation at 2 Hz frequency. The RFA process will be applied to the existing nerves via a generator (TOP Lesion Generator TLG-20, MPS Medical Product Service GmbH, Germany) at 42 C, as pulse RFA for 120 seconds.

To address any discomfort that may occur after the procedure, a total of 2 cc of betamethasone (5 mg+2 mg/1 cc) and %2 lidocaine (1 cc) will be injected into the points where RFA is applied, after aspiration.

For participants who will not be injected at more than 2 points, the same procedure will be applied without activating the generator in order to ensure that the participants remain blind to group allocation and only 2 cc % 0,9 NaCl will be injected into the treatment points. After the procedure, patients will be advised to continue their current medication and exercise therapy. Patients will not receive other pain treatments such as physical therapy, knee re-RFA treatment, intra-articular hyaluronic acid, steroid or similar injection treatments for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30-75
* Chronic knee pain that lasts at least 6 months
* Radiographic confirmation of osteoarthritis: Presence of Grade 3 or 4 radiographic changes characterized by significant narrowing in the medial space of the tibiofemoral joint according to the Kellgren-Lawrence classification system
* Knee pain >40 mm when performing one of the two movements that cause the most severe pain (sitting to standing or going up and down stairs) according to 100 mm VAS

  * 50% reduction in VAS with diagnostic genicular nerve block

Exclusion Criteria:

* Presence of systemic inflammatory disease such as rheumatoid arthritis
* Previous RFA treatment to the knee or hyaluronic acid or steroid injection to the knee within the last 3 months
* History of previous knee surgery
* Clinically significant structural abnormalities other than osteoarthritis that may lead to chronic knee pain
* Having undergone physical therapy to the knee in the last 6 months or a history of knee trauma
* Application of other pain treatments
* Body-Mass İndex <18 and >40 kg/m2
* Pregnancy
* Presence of uncontrolled serious illness (cancer, diabetes, etc.), infection, psychiatric disorder, coagulation disorder

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cybex 770, Humac Norm Dynamometer (CSMI, Stoughton, MA, USA): Isokinetic muscle strength of the quadriceps and hamstring muscles | baseline, 1st month and 3rd month
  Cybex 770, Humac Norm dynamometer (CSMI, Stoughton, MA, USA) will be used to measure the isokinetic muscle strength of the quadriceps and hamstring muscles.
  During the test, while the knee joint moves from 90 degrees to 0 degrees, 5 maximum contraction repetitions are provided at an angular speed of 60/sec for muscle strength and 15 maximum repetitions of contraction at an angular speed of 180/sec are provided for muscle endurance.10-second rest period is left between repetitions.The preparation set is applied before the test.Afterwards, there is a 2-minute rest period before starting the test.Isokinetic knee extensor and flexor mean peak torque is determined and It is standardized according to body weight(Peak torque/body weight:Newton-metre/kg).Higher values in peak torque indicate better levels of muscle strength and endurance.
HUBER 360 Evolution Device (LPG, Valence, France) | baseline, 1st month and 3rd month
  HUBER 360 Evolution device will be used in balance-coordination evoluation.The patient will be placed on a multi-axis platform and 4 different tests will be applied.
Cybex 770, Humac Norm dynamometer (CSMI, Stoughton, MA, USA): Proprioception of the knee joint | baseline, 1st month and 3rd month
  A Cybex 770, Humac Norm dynamometer (CSMI, Stoughton, MA, USA) will be used to measure proprioception of the knee joint. During the test, participants will be blindfolded to eliminate visual input. Initially, for the preparation set, the participants' knee joint will be passively flexed from 90 degrees to 45 degrees and they will be provided with an understanding of the test angle. During the test, the device will enter isokinetic con/con mode and the participant will be able to actively move the knee. When the participant moves the knee to the test angle, the value will be recorded and the absolute angular error, i.e. the difference between the recorded angle and the target angle (45 degrees), will be determined. The test will be repeated 3 times and the values will be averaged.The farther the measured value is from the target value, the more impaired proprioception is.

SECONDARY OUTCOMES:
Romberg Test | baseline, 1st month and 3rd month
  Stability:
  The movement of the patient's center of pressure will be measured with a test inspired by the Romberg test, performed on two feet for 50 seconds with both eyes open and closed.This test evaluates static balance, muscle fatigue, and visual effects.
  In this test, the normal values of the stability coefficient are between 1.11 and 6.77.Values measured outside this range indicate a deterioration in stability.
Single Leg Test | baseline, 1st month and 3rd month
  Single leg test: The balance test on one leg is applied for a maximum of 30 seconds.The right and left side imbalance, that is, the inequality in laterality that affects static balance, determines the risk of falling.The single leg test will be applied to the healthy and diseased sides, and length and area values will be obtained with the test.High length and area values indicate poor balance.
Walking | baseline, 1st month and 3rd month
  This test, which performs stato-dynamic analysis with a vertical ramp for 50 seconds with the arms extended, is inspired by the Fukuda test.It shows the number of steps and is related to walking speed.A minimum of 80 steps must be taken for the test to be evaluated.A high number of steps taken in a fixed time period indicates that the walking speed is at a good level.
Coordination | baseline, 1st month and 3rd month
  It is a test that evaluates the patient's capacity to coordinate movements.During the test, the patient must maintain a constant force in an unstable environment and as quickly as possible.Thus, the capacity to manage multiple tasks simultaneously is evaluated.There are 30 different levels in the test, and the level the patient reaches is determined by the time spent in this process.The difficulty level increases as the level progresses, thus indicating better coordination.
Berg-Balance Test | baseline, 1st month and 3rd month
  It is a test that evaluates the person's performance and determines the balance and risk of falling, and is completed in 15-20 minutes.It consists of 14 general balance activities that change the orientation of the body's center of gravity relative to the support surface and evaluate the ability to maintain a static position during a decrease in the support surface.The patient is evaluated during the activities and each activity is scored on a 5-point scale where the score ranges from 0 to 4.Total score is 56.A score between 0-20 is considered a high risk of falling, a score between 21-40 is considered a medium fall risk, and a score between 41-56 is considered a low fall risk.Changes of 8 points and above indicate that the person's addiction is increasing.
International Falls Efficacy Scale (FES-1) | baseline, 1st month and 3rd month
  The test, which evaluates the fear and anxiety of people about the risk of falling during their daily activities, consists of 16 questions. Each question is scored between 0-4 points. High scores are associated with poor outcomes. It has validity and reliability in Turkish for the older age group.
WOMAC Osteoarthritis Index | baseline, 1st month and 3rd month
  It is a specific, valid, reliable measure recommended by Outcome Measures in Rheumatology Clinical Trials (OMERACT) for osteoarthritis studies. It includes 24 questions in three subgroups: pain, stiffness, and physical function. Each question is scored according to the Likert scale as 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe. The maximum scores that can be obtained from the subgroups are 20 for the pain subgroup, 8 for stiffness, and 68 for physical function. Higher scores indicate increased pain and stiffness and deterioration in physical function.
SF-12 (Short Form-12) | baseline, 1st month and 3rd month
  General quality of life scale: It is a scale that evaluates the impact of health on people's daily lives, which is an abbreviated version of SF-36. It consists of 8 subheadings and a total of 12 questions. 2 subheadings of the scale aim to evaluate physical functionality, 2 physical roles, 1 pain, 1 general health, 1 energy, 1 social functionality, 2 emotional roles and 2 mental health. Physical Component Score (SF-12 P) and Mental Component Score (SF-12 M) can be accessed with online calculation tools. High scores indicate high quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Physical Medicine and Rehabilitation, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Michael JW, Schluter-Brust KU, Eysel P. The epidemiology, etiology, diagnosis, and treatment of osteoarthritis of the knee. Dtsch Arztebl Int. 2010 Mar;107(9):152-62. doi: 10.3238/arztebl.2010.0152. Epub 2010 Mar 5. PMID 20305774
- [Background] Crawford DC, Miller LE, Block JE. Conservative management of symptomatic knee osteoarthritis: a flawed strategy? Orthop Rev (Pavia). 2013 Feb 22;5(1):e2. doi: 10.4081/or.2013.e2. Print 2013 Feb 22. PMID 23705060
- [Background] Williams SB, Brand CA, Hill KD, Hunt SB, Moran H. Feasibility and outcomes of a home-based exercise program on improving balance and gait stability in women with lower-limb osteoarthritis or rheumatoid arthritis: a pilot study. Arch Phys Med Rehabil. 2010 Jan;91(1):106-14. doi: 10.1016/j.apmr.2009.08.150. PMID 20103404
- [Background] Chang AH, Lee SJ, Zhao H, Ren Y, Zhang LQ. Impaired varus-valgus proprioception and neuromuscular stabilization in medial knee osteoarthritis. J Biomech. 2014 Jan 22;47(2):360-6. doi: 10.1016/j.jbiomech.2013.11.024. Epub 2013 Nov 25. PMID 24321442
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Ajrawat P, Radomski L, Bhatia A, Peng P, Nath N, Gandhi R. Radiofrequency Procedures for the Treatment of Symptomatic Knee Osteoarthritis: A Systematic Review. Pain Med. 2020 Feb 1;21(2):333-348. doi: 10.1093/pm/pnz241. PMID 31578561
- [Background] Conger A, Gililland J, Anderson L, Pelt CE, Peters C, McCormick ZL. Genicular Nerve Radiofrequency Ablation for the Treatment of Painful Knee Osteoarthritis: Current Evidence and Future Directions. Pain Med. 2021 Jul 25;22(Suppl 1):S20-S23. doi: 10.1093/pm/pnab129. PMID 34308957
- [Background] Guven Kose S, Kirac Unal Z, Kose HC, Celikel F, Akkaya OT. Ultrasound-guided genicular nerve radiofrequency treatment: prospective randomized comparative trial of a 3-nerve protocol versus a 5-nerve protocol. Pain Med. 2023 Jul 5;24(7):758-767. doi: 10.1093/pm/pnad025. PMID 36869680
- [Background] Chang YW, Tzeng IS, Lee KC, Kao MC. Functional Outcomes and Physical Performance of Knee Osteoarthritis Patients After Ultrasound-Guided Genicular Nerve Radiofrequency Ablation. Pain Med. 2022 Feb 1;23(2):352-361. doi: 10.1093/pm/pnab280. PMID 34534349
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Ulus Y, Durmus D, Akyol Y, Terzi Y, Bilgici A, Kuru O. Reliability and validity of the Turkish version of the Falls Efficacy Scale International (FES-I) in community-dwelling older persons. Arch Gerontol Geriatr. 2012 May-Jun;54(3):429-33. doi: 10.1016/j.archger.2011.06.010. Epub 2011 Aug 9. PMID 21831462
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] Tuzun EH, Eker L, Aytar A, Daskapan A, Bayramoglu M. Acceptability, reliability, validity and responsiveness of the Turkish version of WOMAC osteoarthritis index. Osteoarthritis Cartilage. 2005 Jan;13(1):28-33. doi: 10.1016/j.joca.2004.10.010. PMID 15639634
- [Background] Thomsen MG, Latifi R, Kallemose T, Husted H, Troelsen A. Does knee awareness differ between different knee arthroplasty prostheses? A matched, case-control, cross-sectional study. BMC Musculoskelet Disord. 2016 Apr 1;17:141. doi: 10.1186/s12891-016-1001-3. PMID 27036995
- [Background] Soylu C, Kutuk B. Reliability and Validity of the Turkish Version of SF-12 Health Survey. Turk Psikiyatri Derg. 2022 Summer;33(2):108-117. doi: 10.5080/u25700. English, Turkish. PMID 35730511
- [Background] Shanahan EM, Robinson L, Lyne S, Woodman R, Cai F, Dissanayake K, Paddick K, Cheung G, Voyvodic F. Genicular Nerve Block for Pain Management in Patients With Knee Osteoarthritis: A Randomized Placebo-Controlled Trial. Arthritis Rheumatol. 2023 Feb;75(2):201-209. doi: 10.1002/art.42384. Epub 2022 Nov 11. PMID 36369781
- [Background] Cankurtaran D, Karaahmet OZ, Yildiz SY, Eksioglu E, Dulgeroglu D, Unlu E. Comparing the effectiveness of ultrasound guided versus blind genicular nerve block on pain, muscle strength with isokinetic device, physical function and quality of life in chronic knee osteoarthritis: a prospective randomized controlled study. Korean J Pain. 2020 Jul 1;33(3):258-266. doi: 10.3344/kjp.2020.33.3.258. PMID 32606270